CLINICAL TRIAL: NCT04033679
Title: The Effects of Adjunctive Transcranial Direct Current Stimulation on Treatment Adherence in Schizophrenia
Brief Title: The Effects of Non-invasive Brain Stimulation on Treatment Adherence in Schizophrenia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Philip Gerretsen, Clinicial Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 103-2018
Record Dates: First submitted 2019-05-23; First posted 2019-07-26 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia;Schizoaffective
Keywords: Magnetic resonance imaging; Brain stimulation; Medication adherence
MeSH Terms: conditions — Psychotic Disorders; Medication Adherence

STUDY DESIGN:
Intervention Model Description: Participant randomly assigned to receive either TDCS stimulation or sham stimulation.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active TDCS (Experimental): In the active condition, a constant current of 2 mA intensity will be applied for 20 min to the parietal regions, using P3 as the cathode and P4 as the anode.
  Interventions: Other: Active TDCS
- Sham TDCS (Sham Comparator): In the sham condition, stimulation will be administered using the same parameters at the site of active treatment, but the current will be turned off after 30 seconds.
  Interventions: Other: Sham TDCS

INTERVENTIONS:
Other: Active TDCS — Participants will receive active TDCS stimulation.
  Arms: Active TDCS
Other: Sham TDCS — Participants will receive sham TDCS stimulation.
  Arms: Sham TDCS

SUMMARY:
This study seeks to explore the effects of transcranial direct current stimulation (tDCS), a non-invasive method of brain stimulation, as an adjunctive treatment to improve antipsychotic medication adherence in patients with schizophrenia (SCZ). The investigators hypothesize that 20 sessions of tDCS will improve medication nonadherence in patients with SCZ.

DETAILED DESCRIPTION:
The proposed study will investigate the effects of adjunctive tDCS on antipsychotic medication adherence by targeting brain regions implicated in impaired insight, a primary contributor to medication nonadherence in patients with SCZ. Participants will be randomized to receive either active or sham tDCS. tDCS will be administered twice-daily for 10 days (20 sessions) excluding weekends. Brain scans will be performed before and after 10 days of tDCS. Antipsychotic drug adherence will be assessed based primarily on pill-count, and secondarily, plasma level concentrations and clinician-judgement.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants of any race or ethnicity
2. Inpatients or outpatients ≥18 years of age
3. DSM-V diagnosis of SCZ or schizoaffective disorder
4. Capable of consenting to participate in the research study
5. On a stable dose of antipsychotic drug and other concomitant medications for at least 2 months, and unlikely to undergo changes in dose during the study

Exclusion Criteria:

1. Unwilling or incapable to consent to the study based on the MacArthur Test of Competence
2. Unstable medical or any concomitant major medical or neurological illness, including a history of seizures
3. Acute suicidal or homicidal ideation
4. Formal thought disorder rating ≥3 on the Positive and Negative Syndrome Scale (PANSS) P2 conceptual disorganization item
5. DSM-V substance dependence (except caffeine and nicotine) within 1 month of entering the study*
6. Positive urine drug screen except for cannabis/marijuana at the screening visit
7. Metal implants or pacemaker precluding an MRI scan or other contraindications to MRI (eg., claustrophobia)
8. Pregnancy
9. Score < 32 on the Wide Range Achievement Test-III

   * Substance misuse: In addition to impaired insight, substance misuse is one of the principle contributors to medication nonadherence. To minimize the possibility of its influence, participants with a DSM-V diagnosis of substance dependence within 1 month of entering the study or a positive urine drug test (except for cannabis/marijuana) at the screening visit will be excluded. Substance use and urine drug screens will be assessed at subsequent study visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2019-08-15 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Medication adherence - Pill Count | During 3-month follow up phase
  Pill count or percentage of weekly antipsychotic medication adherence will be assessed during the 3-month follow up phase after TDCS is completed.
Medication adherence - Plasma Monitoring | Blood concentration of antipsychotic medication will be measured on day of the first TDCS session before TDCS starts, after 1 week of TDCS is completed, after 2 weeks of TDCS are completed, and during the 3-month follow up phase.
  Blood concentrations of antipsychotic medication will be measured at different points in the study to assess medication adherence.
Medication adherence - Clinician Rating | During 3-month follow up phase
  The Clinician Adherence Rating Scale is a 7-point clinician rated measure which takes into account patients' self-report, medication adherence, and changes in plasma concentrations to provide a comprehensive assessment of antipsychotic medication adherence. A higher score represents greater adherence.

SECONDARY OUTCOMES:
Insight into Psychosis | Illness awareness will be assessed before the TDCS phase begins, after 2 weeks of TDCS are completed, and during the 3-month follow up period
  Level of illness awareness will be assessed by the VAGUS Insight into Psychosis scale. The VAGUS assesses the core domains of insight into psychosis. VAGUS has both self-report and clinician-rated versions with good inter-scale reliability and test-retest reliability. Higher scores indicate better insight into illness.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Gerretsen, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Centre for Addiction and Mental Health (CAMH) is the leading mental health and addictions research facility in Canada, and one of the largest in the world. — https://www.camh.ca/en/science-and-research